CLINICAL TRIAL: NCT02358213
Title: Evaluation of the Reproducibility Inter-observer of the Ultrasound Anomalies of the Salivary Glands in Sjogren's Disease : Etude ETREINTE.
Brief Title: Evaluation of the Reproducibility Inter-observer of the Ultrasound Anomalies of the Salivary Glands in Sjogren's Disease
Acronym: ETREINTE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double
Other Study IDs: RB 14.133 ETREINTE
Record Dates: First submitted 2015-01-26; First posted 2015-02-06 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-03

CONDITIONS: Sjogren's Disease
Keywords: reproductibility
MeSH Terms: conditions — Sjogren's Syndrome | interventions — High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Procedure (Other): 5 ultrasounds were done on 20 patients by 5 different sonographers
  Interventions: Procedure: Ultrasound

INTERVENTIONS:
Procedure: Ultrasound — Ultrasound examinations are done 5 times

SUMMARY:
This aim of this study is to compare the reproducibility of reading of five international experts concerning the anomalies of the salivary glands.

The reproducibility is measure on patients and not on recorded data.

ELIGIBILITY:
Inclusion Criteria:

* Men and women from 18 to 80 years old
* Patients recruited during the multidisciplinary consultation of Sjogren's Disease, filling the criteria of Sjogren's Disease or patients having a salivary recidivate pathology and selected players on the basis of their voluntary service to benefit from an ultrasound of the main salivary glands
* The patients will have to be capable of adhering to the protocol of study and of having understood it.
* The patients will have to be capable of giving a signed informed consent, the latter being obtained before the inclusion

Exclusion Criteria:

* Not cooperative patient and having refused to sign the informed consent.
* Patient incapable to understand the protocol, under guardianship or under guardianship.
* Unaffiliated patients to the Social Security.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Reproducibility between experts | 1 day
  The outcome measure will be assessed bythe answer of a questionnaire which will be complete by the 5 international experts.

SECONDARY OUTCOMES:
Reproducibility by the sonographer | 1 day
  The sonographer's reproductibility will be assesses by the answer of a questionnaire which will be complete by the 5 international experts.

CONTACTS AND LOCATIONS:
Overall Officials: Valérie DEVAUCHELLE, PUPH, Principal Investigator — Hospital Brest